CLINICAL TRIAL: NCT02937610
Title: Prospective Experience of Percutaneous Endoscopic Gastrostomy Tubes in an Otolaryngologist Service - Safety and Benefits
Brief Title: Percutaneous Endoscopic Gastrostomy in Hands of ORL-HN Surgeon
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Leif Back, MD PhD, University of Helsinki
Other Study IDs: JR/Helsinki/ORL/3
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Head and Neck Cancer; Percutaneous Endoscopic Gastrostomy; Complication
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: percutaneous endoscopic gastrostomy — PEG tube inserted with pull technique
  Other Names: PEG

SUMMARY:
PEG tubes are commonly used to provide nutritional support to patients with head and neck cancer. PEG insertions are typically carried out by gastroenterologists, but also otorhinolaryngologist - head and neck surgeons perform the procedure in some countries. Prospective studies on PEG tube placements in an ORL - HNS service are lacking. The investigators aim was to prospectively evaluate the preformance of ORL - HN surgeons in PEG tube insertions, and analyze the time gains and cost effectiveness achieved of the independency from other specialities.

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer as a underlying disease

Exclusion Criteria:

-

Ages: 31 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 127 consecutive head and neck cancer patients, who underwent PEG placement at the Department of ORL - HNS, Helsinki University Hospital, between October 2011 and May 2013.
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
complications | 1 year
mortality | 1 year

SECONDARY OUTCOMES:
delay | 1 year
  delay from the decision to insert PEG to the procedure

OTHER OUTCOMES:
costs | 1 year
  cost of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Ruohoalho, MD, Principal Investigator — Otorhinolaryngology - Head and Neck Surgery

IPD SHARING:
Plan to Share IPD: No